CLINICAL TRIAL: NCT03934970
Title: A Study of Diffusion Tensor Imaging of Median Nerve in Diabetic Peripheral Neuropathy
Brief Title: Diffusion Tensor Imaging of Median Nerve in Diabetic Peripheral Neuropathy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelalim, Clinial Professor of Neurology, Cairo University
Other Study IDs: 19/04/15
Record Dates: First submitted 2019-01-26; First posted 2019-05-02 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Diabetic Polyneuropathy; Magnetic Resonance Imaging
Keywords: Diabetic Polyneuropathy; Diffusion tensor imaging; Neuropathy scores
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic Neuropathy: Thirty Egyptian patients with type 2 diabetes mellitus complaining of symptoms suggestive of peripheral neuropathy including 12 males and 18 females with a mean of 50.90 ± 9.18.
  Interventions: Diagnostic Test: Diffusion tensor imaging of peripheral nerves
- Healthy Control Subjects: Fifteen normal healthy Egyptian volunteers including10 males and 5 females with a mean age of 45.67±7.77 years.
  Interventions: Diagnostic Test: Diffusion tensor imaging of peripheral nerves

INTERVENTIONS:
Diagnostic Test: Diffusion tensor imaging of peripheral nerves — All subjects underwent evaluation using 1.5T DTI of median nerves and NCS. Patients underwent clinical evaluation using Neuropathy Deficit Score (NDS), Neuropathy Impairment Score in the Lower Limbs (NIS-LL) and Diabetic Neuropathy Examination (DNE) score.
  Other Names: Nerve conduction studies; Neuropathy clinical scores

SUMMARY:
This study is a diagnostic accuracy study that aims to evaluate the role of DTI in evaluation of DPN in comparison to clinical scores and nerve conduction studies (NCS). The study included 30 patients with diabetes mellitus complaining of neuropathy symptoms and 15 healthy volunteers. All subjects underwent evaluation using 1.5T DTI of median nerves and NCS. Patients underwent clinical evaluation using Neuropathy Deficit Score (NDS), Neuropathy Impairment Score in the Lower Limbs (NIS-LL) and Diabetic Neuropathy Examination (DNE) score. The values of these tests were compared and correlated and diagnostic accuracy tests were performed together with identification of cut-off score for abnormal diffusion tensor imaging parameters in diabetic neuropathy

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with symptoms suggestive of peripheral neuropathy.

Exclusion Criteria:

* Patients with evidence of nerve entrapment or neuropathy due to causes other than DM

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a case-control study of 30 Egyptian patients with type 2 diabetes mellitus complaining of symptoms suggestive of peripheral neuropathy including 12 males and 18 females with a mean of 50.90 ± 9.18 years and 15 normal healthy Egyptian volunteers including10 males and 5 females with a mean age of 45.67±7.77 years.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Comparison of diagnostic accuracy of Diffusion tensor imaging in comparison to nerve conduction velocity | Six Months
  This is a diagnostic accuracy study comparing the ability of Diffusion Tensor Imaging to diagnose Diabetic neuropathy. This is performed in comparison to nerve conduction studies which is a well established quantitative and qualitative diagnostic test that measures nerve conduction velocity in meter/second.
Comparison of diagnostic accuracy of Diffusion tensor imaging of peripheral nerves in comparison to motor amplitude in diabetic patients. | Six Months
  This is a diagnostic accuracy study comparing the ability of Diffusion Tensor Imaging to diagnose Diabetic neuropathy. This is performed in comparison to nerve conduction studies which is a well established quantitative and qualitative diagnostic test that measures motor amplitude in millivolt.
Comparison of diagnostic accuracy of Diffusion tensor imaging of peripheral nerves in comparison to sensory amplitude in diabetic patients. | Six Months
  This is a diagnostic accuracy study comparing the ability of Diffusion Tensor Imaging to diagnose Diabetic neuropathy. This is performed in comparison to nerve conduction studies which is a well established quantitative and qualitative diagnostic test that measures sensory amplitude in microvolt.
Comparison of diagnostic accuracy of Diffusion tensor imaging of peripheral nerves in comparison to Neuropathy Deficit Score in diabetic patients. | Six Months
  This is a diagnostic accuracy study comparing the ability of Diffusion Tensor Imaging to diagnose Diabetic neuropathy in comparison to Neuropathy Deficit Score which examines vibration, sensation (0 if present and normal and 1 if absent reduced or uncertain) and ankle reflex (0 if present and normal, and 2 if absent) with a maximum total score of 10. The grades of severity are mild (3-5) moderate (6-8) and severe (9-10).
Comparison of diagnostic accuracy of Diffusion tensor imaging of peripheral nerves in comparison to Neuropathy Impairment Score in diabetic patients. | Six Months
  This is a diagnostic accuracy study comparing the ability of Diffusion Tensor Imaging to diagnose Diabetic neuropathy in comparison to Neuropathy Impairment Score in the Lower Limbs which evaluates the changes in motor, sensory and reflex activity. The scale ranges from the normal value at "0" points, with a maximum value of 88 points.
Comparison of diagnostic accuracy of Diffusion tensor imaging of peripheral nerves in comparison to Diabetic Neuropathy Examination in diabetic patients. | Six Months
  This is a diagnostic accuracy study comparing the ability of Diffusion Tensor Imaging to diagnose Diabetic neuropathy in comparison to Diabetic Neuropathy Examination score which tests only the limbs of right side with a maximum score of 16 points. A score, greater than three, is considered abnormal.

SECONDARY OUTCOMES:
Identifying cut-off value for abnormal diffusion tensor fractional anisotropy in diabetic neuropathy. | Six months
  This study aims to identify cut-off absolute value of fractional anisotropy that is considered abnormal in diabetic neuropathy. Fractional anisotropy (FA) is a scalar value between zero and one that describes the degree of anisotropy of a diffusion process. A value of zero means that diffusion is isotropic, i.e. it is unrestricted (or equally restricted) in all directions. A value of one means that diffusion occurs only along one axis and is fully restricted along all other directions.
Identifying cut-off value for abnormal diffusion tensor apparent diffusion coefficient in diabetic neuropathy. | Six months
  This study aims to identify cut-off absolute value of apparent diffusion coefficient (ADC) that is considered abnormal in diabetic neuropathy. An ADC of a tissue is expressed in units of mm2/s. There is no unanimity regarding the boundaries of the range of normal diffusion, but ADC values less than 1.0 to 1.1 x 10-3 mm2/s (or 1000-1100 x 10-6 mm2/s) are generally acknowledged in adults as indicating restriction.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelalim, MD, Principal Investigator — Department of Neurology, Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No